CLINICAL TRIAL: NCT00410644
Title: A Repeated-Dose Evaluation of Analgesic Use and Safety of Dilaudid SR (Hydromorphone HCI) in Patients With Chronic Non-Malignant Pain
Brief Title: A Repeated-Dose Evaluation of a Pain Relieving Drug Use and Safety of OROS Hydromorphone HCI in Patients With Chronic Non-Malignant Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CR011617
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Pain; Analgesics; Opioid
Keywords: Non-malignant chronic pain; pain; analgesics; opioid
MeSH Terms: conditions — Pain

INTERVENTIONS:
Drug: OROS Hydromorphone HCI

SUMMARY:
The purpose of this repeated dose study is to develop recommended dosing information for initiation of therapy with OROS Hydromorphone in patients with chronic non-malignant pain converting from other strong oral or transdermal opioids. It will also assist in the development of a recommended starting dose by which patients can be titrated to an appropriate maintenance dose of OROS Hydromorphone HCI. The safety profile for OROS Hydromorphone HCI will also be evaluated.

DETAILED DESCRIPTION:
This single-blind (with respect to dose), repeated dose study evaluating patients with chronic non-malignant pain was conducted in tandem with a similar protocol in patients with chronic cancer pain. A total of 463 patients were enrolled and evaluated in these studies. Patients receiving chronic opioid therapy were converted to once daily OROS hydromorphone using oral morphine equivalents. Supplementary immediate-release (IR) hydromorphone was provided for breakthrough pain. The dose of OROS hydromorphone was escalated after every 2 days of therapy until no more than 3 doses of immediate-release(IR) hydromorphone were required in a 24-hour period. Once a patient could be maintained on a stable dose of OROS hydromorphone for 3 consecutive days, the patient entered a 2-week maintenance phase. Patients who completed the study were eligible for participation in an OROS hydromorphone long-term extension study, Study DO-109. The hypothesis is the 24-hour controlled-release form of oral hydromorphone may provide consistent pain relief, convenient dosing, and enhanced compliance while possibly decreasing the incidence of side effects associated with peak (high) and trough (low) fluctuations in plasma drug concentrations typically seen with immediate-release dosage formulations. Patients received OROS Hydromorphone HCI at Visit 2,3, and 4(either 8,16,32, and/or 64mg tablets) taken orally. OROS Hydromorphone HCI doses were titrated after every two days of therapy as necessary until dose stabilization occurred, followed by a two week Maintenance Therapy Phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have chronic non-malignant pain, including pain associated with AIDS, who are currently receiving strong oral or transdermal opioid analgesics, or patients who are currently receiving opioids plus non-opioid combination analgesics, and have persisting pain
* patients who require at least 45 mg of oral morphine or opioid equivalent every 24 hours for the management of chronic non-malignant pain
* patients who can reasonably be expected to have stable opioid requirements for the duration of the study.

Exclusion Criteria:

* Patients intolerant of or hypersensitive to hydromorphone (or other opioid agonists)
* patients who have dysphagia or are unable to swallow tablets
* patients who are pregnant or breast-feeding
* patients with severe respiratory compromise or severely depressed ventilatory function
* patients with any gastrointestinal disorder, including pre-existing severe GI narrowing(pathologic or iatrogenic), that may affect the absorption or transit of orally administered drugs or have an acute abdominal condition that may be obscured by opioids
* patients with clinically significant impaired renal or hepatic function, Addison's disease, hypothyroidism, prostatic hypertrophy, or urethral stricture
* patients who are known active drug abusers or alcoholics
* patients with any significant CNS disorder, including but not limited to head injury, intracranial lesion, increased intracranial pressure, seizure disorder, stroke within the past 6 months, and disorders of cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Study Completion 1999-02 (Actual)

PRIMARY OUTCOMES:
No primary efficacy variable was defined in report. Protocol variables measured included: Total daily dose of OROS hydromorphone, daily use of rescue medication, daily pain relief scores, and time/number of steps needed for dose stabilization.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- [Derived] Wallace M, Rauck RL, Moulin D, Thipphawong J, Khanna S, Tudor IC. Conversion from standard opioid therapy to once-daily oral extended-release hydromorphone in patients with chronic cancer pain. J Int Med Res. 2008 Mar-Apr;36(2):343-52. doi: 10.1177/147323000803600218. PMID 18380946
- [Derived] Wallace M, Rauck RL, Moulin D, Thipphawong J, Khanna S, Tudor IC. Once-daily OROS hydromorphone for the management of chronic nonmalignant pain: a dose-conversion and titration study. Int J Clin Pract. 2007 Oct;61(10):1671-6. doi: 10.1111/j.1742-1241.2007.01500.x. PMID 17877652